CLINICAL TRIAL: NCT00581659
Title: Evaluation of the Bausch & Lomb PureVision Under Nighttime Driving Conditions
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Timothy L. Brown, Associate Research Scientist, University of Iowa
Other Study IDs: 200709761
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lens A, Lens B: The first independent variable is the contact lens. Each subject will wear both PureVision (TM0 aspheric contact lenses and conventional spherical contact lenses on separate visits. The second independent variable is visibility condition. Subjects will complete the study drive both in clear nighttime conditions and at night under glare conditions. In both cases, the driver will experience oncoming traffic; however, in the glare condition, the simulator will be equipped with a point light source sufficient to provide glare similar to that provided by oncoming traffic in the real world.

SUMMARY:
The objective of this study is to quantify differences in nighttime driving performance between the Bausch & Lomb PureVision™ aspheric contact lenses and a conventional spherical contact lens.

The primary aims of this study are to determine the differences between B&L PureVision™ aspheric contact lenses and a conventional spherical contact lens in visual performance measures associated with driving, such as number of objects seen.

The secondary aims of this study are to determine differences between B&L PureVision™ aspheric contact lenses and a conventional spherical contact lens in driving performance measures such as number of objects hit.

DETAILED DESCRIPTION:
Contact lenses have the potential to affect visual performance in various driving situations, including low-visibility situations such as driving at night. This study will assess the effect on typical nighttime driving tasks such as reading signs and avoiding road hazards.

This is a single-site study. Individuals who are currently spherical contact lens wearers, who believe they have little or no astigmatism, and who are licensed drivers will be invited to partipate in this study. Twenty-four completed subjects are required. This study will involve a 2x2 within-subject comparison.

The first independent variable is the contact lens. Each subject will wear both PureVision (TM0 aspheric contact lenses and conventional spherical contact lenses on separate visits. The second independent variable is visibility condition. Subjects will complete the study drive both in clear nighttime conditions and at night under glare conditions. In both cases, the driver will experience oncoming traffic; however, in the glare condition, the simulator will be equipped with a point light source sufficient to provide glare similar to that provided by oncoming traffic in the real world.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

* valid US driver's license
* drive at least 100 miles per month
* not restricted to driving at night
* willing to travel to the National Advanced Driving Simulator
* currently successfully wear soft spherical contact lenses
* between the ages of 25 and 45
* no previous participation in any vision simulator driving studies

Exclusion Criteria:

Exclusion Criteria

* known or suspected pregnancy
* current serious illness or have received radiation and/or chemotherapy treatment within the last 6 months
* Type 1 Diabetics or Untreated Type II Diabetics
* current heart condition or heart attack, or pacemaker implanted within last 6 months
* known seizure disorder or epilepsy
* Meniere's disease or any inner ear, vertigo, hearing, or balance conditions
* known narcolepsy
* Chronic Fatigue Syndrome
* untreated sleep apnea
* uncontrolled asthma or chronic bronchitis
* Chronic Obstructive Pulmonary Disease
* migraine headaches that require narcotic medications
* untreated depression or anxiety disorder
* claustrophobia
* drug dependency
* untreated ADHD
* taking current prescription or over-the-counter medications that create sedation or drowsiness
* uncontrolled glaucoma or glaucoma under current treatment
* propensity toward motion sickness
* new diagnosis of dementia by physician
* diagnosis of macular degeneration
* experience any side effects from dilation of the eyes
* Diabetes-induced eye disease in either eye
* Cataract surgery in either eye or currently have cataracts
* refractive eye surgery in either eye
* more than 0.25 diopters of refractive astigmatism in either eye
* less than 0.05 microns of positive spherical aberration in either eye -refractive error less than -0.50 diopters or greater than -3.00 diopters -

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects who currently wear spherical contact lenses and believe they have little or no astigmatism and are licensed drivers.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint measured is the number of objects on the roadway that were detected - a count of the total number of objects that the driver correctly detects out of the total number of objects present. | at time of both drives

SECONDARY OUTCOMES:
The secondary aims of this study are to determine differences between B&L PureVision™ aspheric contact lenses and a conventional spherical contact lens in driving performance measures such as number of objects hit. | at the time of both drives

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wilkinson, OD, Principal Investigator — National Advanced Driving Simulator
Locations (1):
- National Advanced Driving Simulator, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared